CLINICAL TRIAL: NCT06326203
Title: Randomized, Prospective, Controlled, Single-center, Open-label Phase II Clinical Trial Aimed at Evaluating the Safety and Efficacy of Autologous Mesenchymal Stem Cell Therapy for Lower Limb Ulcers in Patients With Critical Limb Ischemia
Brief Title: Cell Therapy for Lower Limb Ulcers in Patients With Critical Limb Ischemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Matheus Bertanha, PhD, Professor, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPECLIN-MB-8
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Arterial Disease; Leg Ulcer
MeSH Terms: conditions — Peripheral Arterial Disease; Leg Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMBRYONIC STEM CELLS (Experimental): Cellular Therapy Treatment: The treatment will consist of **20 participants (n=20) who will receive treatment with expanded mesenchymal stem cells (MSCs). The patient will undergo a surgical debridement procedure for the ulcer to be in its optimal condition (Visit 1). Subsequently, the patient will receive MSC application via perilesional injections and a biocovering produced by the study team, also containing the same cells (single session - the MSC-containing dressing will remain in contact with the ulcer for 7 days). After removal of the biological dressing, the ulcer will receive local care with a topical hydrogel dressing, dry gauze, and a crepe bandage, with a minimum of one change per day.
  Interventions: Biological: CELULAS TRONCO
- CONVENTIONAL DRESSING (Control Group) (Active Comparator): The control group will consist of 20 participants (n=20) who will receive local care for the ulcer. The patient will undergo a surgical debridement procedure for the ulcer to be in its optimal condition (Visit 1). Subsequently, the patient will receive the application of a conventional dressing with Hydrogel, dry gauze, and a crepe bandage. The patient will be instructed to change the dressing at least once a day.
  Interventions: Device: CONVENTIONAL DRESSING

INTERVENTIONS:
Biological: CELULAS TRONCO — Cellular Therapy Treatment: The treatment will consist of **20 participants (n=20) who will receive treatment with expanded mesenchymal stem cells (MSCs). The patient will undergo a surgical debridement procedure for the ulcer to be in its optimal condition (Visit 1). Subsequently, the patient will receive MSC application via perilesional injections and a biocovering produced by the study team, also containing the same cells (single session - the MSC-containing dressing will remain in contact with the ulcer for 7 days). After removal of the biological dressing, the ulcer will receive local care with a topical hydrogel dressing, dry gauze, and a crepe bandage, with a minimum of one change per day.
  Arms: EMBRYONIC STEM CELLS
Device: CONVENTIONAL DRESSING — The control group will consist of 20 participants (n=20) who will receive local care for the ulcer. The patient will undergo a surgical debridement procedure for the ulcer to be in its optimal condition (Visit 1). Subsequently, the patient will receive the application of a conventional dressing with Hydrogel, dry gauze, and a crepe bandage. The patient will be instructed to change the dressing at least once a day.
  Arms: CONVENTIONAL DRESSING (Control Group)

SUMMARY:
Peripheral arterial disease (PAD) can progress to critical limb ischemia (CLI) of the affected lower limb, characterized by pain at rest, ulcerations or gangrene, with a high risk of amputation. In this phase, the best treatment is arterial limb revascularization, but this is not always possible or even effective for promoting pain relief, healing of ulcers or preventing amputations, in addition to the high socioeconomic cost caused by the disease. Recent advances in cell therapy represent a promising supporting alternative for the treatment of PAD in cases where conventional alternatives have run out. Objective: To evaluate the safety and efficacy of cell therapy with expanded autologous mesenchymal stem cells in the treatment of patients with PAD with CLI and chronic arterial ulcers. Methods: An open randomized clinical study will be performed with 2 groups of 20 patients with CLI: in group 1, a fragment of abdominal fat tissue (10g) will be collected to obtain mesenchymal stem cells, which will be expanded and applied using subcutaneous perilesional injection in the affected lower limb, in addition to the application in the form of a personalized curative biological on the wounds. Group 2 will receive conventional treatment with a Hydrogel dressing with essential fatty acids. Periodic clinical evaluations, complementary exams and photographic record will be carried out. The main outcome of effectiveness will be partial or total wound healing. Safety outcomes will be monitored for infections, gangrene, amputations and deaths. Participants will be monitored for 120 days. Major amputation cases will not be included. An independent external evaluator and blind to the groups will evaluate the results. It is an innovative procedure with high impact and financial return for SUS, in view of the high prevalence of the disease and the high socioeconomic impact of the disease when it progresses to limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* Absence of distal pulses in the leg (anterior tibial and posterior tibial) and presence or absence of popliteal pulse.
* Peripheral Arterial Disease (PAD).
* Having foot or leg ulcer(s) (distal third) with a minimum area of 1cm2 and a maximum of 3 ulcers totaling up to 20cm2 in the lower limb.
* Having previously received conventional dressing treatment for ulcer indicating no improvement over a minimum period of 3 weeks (antibiotic therapy - if necessary - local care such as mechanical, surgical or chemical debridements - if necessary, dressings).
* PAD with IC classified as Fontaine IV and Rutherford 5.
* Having Ankle Brachial Index (ABI) <0.9 in infragenicular arteries (anterior tibial, posterior tibial, and fibular) or ABI>1.3 in one or more infragenicular arteries when suffering from chronic DMT2 (disease duration > 5 years) not subjected to revascularization treatment or subjected to partial revascularization treatment or treatment failure (stenosis or occlusion) in the last 12 months.
* Inability to revascularize the affected limb (do not have visible infragenicular arteries for surgical approach) and or incomplete revascularization of this limb (undergone endovascular and or surgical treatment that was not able to restore infragenicular pulses) and defined by the doctor that the best available treatment from the surgical vascular point of view has already been performed and was not successful in promoting ulcer healing.
* Drug treatment for PAD and for comorbidities.
* Availability to attend medical appointments.

Exclusion criteria:

* Being pregnant or in the puerperium.
* Having a healed ulcer during the screening period.
* Having signs of systemic infection or active infection in the arterial ulcer or infection of surgical prostheses (bypass, pins, screws). They may be eligible again if they have been successfully treated with antibiotics and the infectious focus has been removed.
* Having an ulcer with devitalized tissue (necrosis). They may be eligible again if they have undergone successful surgical debridement or minor amputations (amputation of toes or limited to the forefoot).
* Having neoplasia and/or being in chemotherapy or radiotherapy treatment or in remission for less than 6 months.
* Being on colchicine or immunomodulators.
* Having infectious diseases such as Human Immunodeficiency Virus (HIV), Hepatitis B and C viruses, Human T-cell Lymphotropic Virus (HTLV); due to the risk of contagion during the manipulation of biological material in the laboratory.
* Having undergone amputation at the level of the leg or thigh in the limb intended to be studied.
* Having COVID-19, diagnosed less than 4 weeks ago.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Amputation | 120 days
  Defined by total number of patients subjected to amputation at the knee or tight level.
Ulcer Healing | 7, 30, 60, 90 and 120 days
  Defined by total or partial epithelization of the ulcer as measured in total square centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J de Oliveira Filho, M.D., Principal Investigator — São Paulo State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira Filho FJ, Rodrigues LDS, Amaral SMBD, Mellucci Filho PL, Medolago NB, de Carvalho Bovolato AL, Alvarado RC, Bertanha M. Study protocol for a randomized clinical trial evaluating the safety and efficacy of autologous adipose-derived stem cell therapy for ulcers in patients with critical limb ischemia. PLoS One. 2025 Apr 9;20(4):e0318922. doi: 10.1371/journal.pone.0318922. eCollection 2025. PMID 40202953